CLINICAL TRIAL: NCT07312344
Title: Exploring the Impact of Exercise-derived Extracellular Vesicle in Blood and Physical Fitness Data in Overweight/Obesity Individuals on Lymphangiogenesis
Brief Title: Impact of Exercise-derived Extracellular Vesicle in Blood and Physical Fitness Data in Overweight/Obesity Individuals
Acronym: Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MURA2025/678; 2025/1365 (Registry Identifier: Mahidol University Multi-faculty Cooperative IRB Review)
Record Dates: First submitted 2025-11-30; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: Exercise; obesity; extracellular vesicle; clinical assessment; physical fitness
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-intensity interval training exercise (Experimental): High-intensity interval training exercise 3 days per week for 6 weeks
  Interventions: Device: High-intensity interval training exercise on treadmill

INTERVENTIONS:
Device: High-intensity interval training exercise on treadmill — High-intensity interval training exercise using 65% to 80% of heart rate max
  Other Names: HIIT; treadmill running

SUMMARY:
This project aims to study the effect of exercise in the obesity/overweight on the changes of physical fitness and blood components. This will provide novel knowledge for medical staffs, researchers, or companies developing alternative strategies for treating obesity/overweight, including drug development and health promotion project to delay or prevent the onset of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged between 25-45 years
2. Thai nationality
3. Ability to walk or perform daily activities independently, without the use of an assistive device
4. Body mass index (BMI) between 25-35 kg/m²
5. Low physical activity levels or sedentary lifestyle based on the World Health Organization 2020

   * The levels of moderate-intensity physical activity < 150-300 minutes per week or the levels of vigorous-intensity physical activity < 75-150 minutes per week
   * Moderate-intensity physical activity: fast walking and bicycling. Vigorous-intensity physical activity: running, aerobic dance, and swimming All participants are required to meet all inclusion criteria to be eligible for the research project.

Exclusion Criteria:

1. Smoking, substance abuse, or alcohol addiction
2. History of respiratory diseases, such as asthma, emphysema, or chronic obstructive pulmonary disease
3. History of cardiovascular diseases, such as coronary heart disease, aortic disease, arrhythmia, or deep vein thrombosis
4. History of high blood pressure (hypertension)
5. History of vestibular system diseases, such as Meniere's disease or otitis media
6. History of neurological disease, such as severe Parkinson's disease or stroke
7. History of previous lower limb surgery, such as hip, knee, or ankle replacement
8. History of musculoskeletal diseases, such as severe osteoarthritis
9. History of severe brain disease, such as dementia
10. Severe visual or hearing impairment
11. Have a cognitive and comprehensive impairment and unable to complete the intervention
12. Have high physical activity or regularly exercise

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Blood component assessment | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program within 1 hour)
  Participant's blood components, e.g. extracellular vesicles, will be investigated by cell assays and proteomic analysis
Foot pressure distribution | 8 times: Day 1 (Before and after HIIT program), Day 4-7 (after HIIT program only), Day 18 (Before and after HIIT program)
  Foot pressure distribution will be measured using a treadmill (Zebris FDM-T Treadmill System, zebris Medical GmbH, Germany)
Facial and abdominal fat thickness measurement | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Facial and abdominal fat thickness and characteristics will be pictured and analyzed using ultrasound imaging
VO2max | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  VO2max parameter (ml/kg/min) will be examined using Cardio Pulmonary Exercise Test
Body composition | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Body composition (%) will be measured by bioelectrical impedance analysis.
Heart rate | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Heart rate (beat/min) will be measured by pulse oximeters
Grip strength | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Grip strength (kg) will be measured by hand grip dynamometer
Leg strength | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Leg strength (kg) will be measured by back-leg-chest dynamometer
Body weight | Pre-training (Day 1 before HIIT program) and post-training (Day 18 after HIIT program)
  Body weight (kg) will be measured by weighing scale
Body height | Pre-training (Day 1 before HIIT program)
  Body height (cm) will be measured by stadiometer

CONTACTS AND LOCATIONS:
Locations (1):
- Chakri Naruebodindra Medical Institute, Faculty of Medicine Ramathibodi Hospital, Mueang Samut Prakan, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gremeaux V, Drigny J, Nigam A, Juneau M, Guilbeault V, Latour E, Gayda M. Long-term lifestyle intervention with optimized high-intensity interval training improves body composition, cardiometabolic risk, and exercise parameters in patients with abdominal obesity. Am J Phys Med Rehabil. 2012 Nov;91(11):941-50. doi: 10.1097/PHM.0b013e3182643ce0. PMID 22854902
- [Background] Ryan BJ, Schleh MW, Ahn C, Ludzki AC, Gillen JB, Varshney P, Van Pelt DW, Pitchford LM, Chenevert TL, Gioscia-Ryan RA, Howton SM, Rode T, Hummel SL, Burant CF, Little JP, Horowitz JF. Moderate-Intensity Exercise and High-Intensity Interval Training Affect Insulin Sensitivity Similarly in Obese Adults. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2941-59. doi: 10.1210/clinem/dgaa345. PMID 32492705
- [Background] Turk Y, Theel W, Kasteleyn MJ, Franssen FME, Hiemstra PS, Rudolphus A, Taube C, Braunstahl GJ. High intensity training in obesity: a Meta-analysis. Obes Sci Pract. 2017 May 29;3(3):258-271. doi: 10.1002/osp4.109. eCollection 2017 Sep. PMID 29071102
- [Background] He XF, Liu DX, Zhang Q, Liang FY, Dai GY, Zeng JS, Pei Z, Xu GQ, Lan Y. Voluntary Exercise Promotes Glymphatic Clearance of Amyloid Beta and Reduces the Activation of Astrocytes and Microglia in Aged Mice. Front Mol Neurosci. 2017 May 19;10:144. doi: 10.3389/fnmol.2017.00144. eCollection 2017. PMID 28579942
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718
- [Background] Louveau A, Smirnov I, Keyes TJ, Eccles JD, Rouhani SJ, Peske JD, Derecki NC, Castle D, Mandell JW, Lee KS, Harris TH, Kipnis J. Structural and functional features of central nervous system lymphatic vessels. Nature. 2015 Jul 16;523(7560):337-41. doi: 10.1038/nature14432. Epub 2015 Jun 1. PMID 26030524
- [Background] Secker GA, Harvey NL. VEGFR signaling during lymphatic vascular development: From progenitor cells to functional vessels. Dev Dyn. 2015 Mar;244(3):323-31. doi: 10.1002/dvdy.24227. Epub 2014 Dec 4. PMID 25399804